CLINICAL TRIAL: NCT06738771
Title: Antimicrobial Therapy for Infections Due to Pseudomonas Aeruginosa With Difficult-to-treat Resistance: a Real-world, Prospective, Multicenter Cohort Study
Brief Title: Antimicrobial Therapy for Difficult-to-treat Pseudomonas Aeruginosa
Acronym: ADDICT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-HORS RIPH-11
Record Dates: First submitted 2024-11-26; First posted 2024-12-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pseudomonas Infections; Pseudomonas Aeruginosa; Prognosis; Drug Resistance, Multiple, Bacterial; Antibacterial Agents; Beta-lactam Antibiotics
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — DTR P. aeruginosa isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patients with invasive P. aeruginosa DTR infection requiring definitive intravenous antibiotic therapy

SUMMARY:
The primary objective of the ADDICT study is to assess and compare the clinical efficacy of available options for antimicrobial therapy (new beta-lactam/beta-lactamase inhibitor combination, cefiderocol or older agents such as aminoglycosides and colistin) in unselected patients with infection due to difficult-to-treat P. aeruginosa.

DETAILED DESCRIPTION:
Infections due to Pseudomonas aeruginosa isolates with acquired resistances to all first-line antipseudomonal beta-lactams and fluoroquinolones (difficult-to-treat isolates - DTR), pose serious therapeutical challenges, especially in critically ill and/or immunocompromised patients. Certain new beta-lactam/beta-lactamase inhibitor combinations (BL/BLI (beta lactamine/ beta lactamase inhibitor) - i.e., ceftolozane-tazobactam, ceftazidime-avibactam, imipenem-relebactam, others) and cefiderocol have shown promising results for the treatment of infections due to DTR P. aeruginosa. However, multicenter data on their real-life utilization in this indication are still scarce.

The ADDICT study is a prospective, multicenter cohort study including unselected patients with DTR P. aeruginosa infection requiring definite intravenous antimicrobial therapy. The primary objective of the study is to investigate the clinical efficacy of available options (new BL/BLI, cefiderocol or older agents such as aminoglycosides and colistin) in this population. Secondary objectives are to compare the clinical and microbiological efficacy of available options in infections due to DTR P. aeruginosa with in vitro susceptibility to more than one last-resort drug, to compare the incidence of non-ecological adverse events observed with these drugs, to assess the incidence of resistance emergence under therapy and to elucidate the molecular mechanisms of resistance emergence, to assess the benefits and risks of combination therapy in this indication, to compare the acquisition rates of multidrug-resistant bacteria other than DTR P. aeruginosa, and Clostridioides difficile infection, to compare Day-28 and in-hospital all-cause mortality rates.

Patients will be recruited in 60 hospital centers contributing to four French networks of research in infectious diseases and critical care (CRICS-TRIGGERSEP, ReaRezo, OutcomeRéa, RENARCI - PROMISE metanetwork). Clinical variables will be collected through an electronic case-report form. DTR P. aeruginosa isolates will be sent to the National Reference Center of Antimicrobial Resistance in P. aeruginosa for centralized analyses (extended antimicrobial susceptibility testing, MLST, whole-genome sequencing of successive isolates if resistance emergence under therapy).

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or over and requiring intravenous definite antimicrobial therapy for a DTR P. aeruginosa infection

Exclusion Criteria:

* Cystic fibrosis
* P. aeruginosa DTR colonization or P. aeruginosa DTR infection not requiring definitive intravenous antibiotic therapy
* Protected person (under guardianship or curatorship)
* Persons under court protection
* Persons deprived of liberty
* Opposition expressed for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective multicenter cohort
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | Test of cure visit
  Clinical responses will be assessed by local investigators. Clinical cure will be defined as a composite endpoint of survival with no relapse occurring since the end of definite therapy and the complete resolution of all initial clinical signs of infection at the ToC visit (all-cause deaths at the ToC visit will be considered as clinical failures).
Clinical cure | Day 7±2 after the completion of definite therapy
  Clinical responses will be assessed by local investigators. Clinical cure will be defined as a composite endpoint of survival with no relapse occurring since the end of definite therapy and the complete resolution of all initial clinical signs of infection at the ToC visit (all-cause deaths at the ToC visit will be considered as clinical failures).

SECONDARY OUTCOMES:
Microbiological eradication | Day 7
  Negativation of cultures for DTR P. aeruginosa in participants with at least one collected follow-up bacteriological sample (when clinically indicated) before the ToC visit
Resistance emergence | Up to hospital discharge, an average of 1 month
  Any culture growing a DTR P. aeruginosa isolate with resistance to at least one new antimicrobial agent (compared to the first isolate) between the second day of definite therapy and hospital discharge
Non-ecological adverse events | At test-of-cure visit, 7±2 days after the completion of definite therapy
  Any toxicity or allergic reaction attributed to the antimicrobial agent by the local investigator
Non-ecological adverse events | From the first day of definite therapy to the ToC visit
  Any toxicity or allergic reaction attributed to the antimicrobial agent by the local investigator
Acquisition of multidrug-resistant bacteria other than DTR P. aeruginosa | Up to hospital discharge, an average of 1 month
  Culture of any clinical or surveillance sample growing a multidrug-resistant bacteria other than P. aeruginosa
Clostridioides difficile infection | Up to hospital discharge, an average of 1 month
  Documented C. difficile infection
In-hospital death | Up to hospital discharge, an average of 1 month
  All-cause death
Death at Day 28 | Day 28
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Francois BARBIER, Professor, Principal Investigator — Centre Hospitalier Universitaire d'Orléans
Locations (48):
- France (47):
  - CHU Amiens, Amiens
  - CH Argenteuil, Argenteuil
  - CH Bayonne, Bayonne
  - CHU de BESANCON, Besançon
  - CH Bethune, Béthune
  - CHU Avicenne, Bobigny
  - CH Bourgoin-Jallieu, Bourgoin
  - CH Métropole Savoie, Chambéry
  - Ch de Chartres, Chartres
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHI Créteil, Créteil
  - CHU Henri Mondor, Créteil
  - CHI Elbeuf Louviers, Elbeuf
  - CH Sud Essone, Étampes
  - Hopital Raymond Poincaré, Garches
  - CHU Grenoble, Grenoble
  - CH Haguenau, Haguenau
  - CHD Vendée, La Roche-sur-Yon
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CHU Limoges, Limoges
  - CHU Lyon Sud, Lyon
  - CHU Lyon, Lyon
  - CHY Lyon, Lyon
  - Hopital Saint-Joseph Saint Luc, Lyon
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - Chu de Nantes, Nantes
  - CHU de Nice, Nice
  - Centre Hospitalier Universitaire d'Orléans, Orléans
  - Hopital Bichat, Paris
  - Hopital Cochin, Paris
  - Hopital LARIBOISIERE, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopital Saint-Antoine, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint-Louis, Paris
  - CH PAU, Pau
  - CH Perpignan, Perpignan
  - Centre Hospitalier de Périgueux, Périgueux
  - CHU Reims, Reims
  - CH Saint-Lô, Saint-Lô
  - CHRU Strasbourg Haute Pierre, Strasbourg
  - CHU Strasbourg, Strasbourg
  - Hopital Foch, Suresnes
  - CH Tourcoing, Tourcoing
  - CH Vannes, Vannes
  - Hôpital Nord-Ouest de Villefranche sur Saone, Villefranche-sur-Saône
- CHU La Réunion, Saint-Denis, Reunion

REFERENCES:
- [Background] Tamma PD, Aitken SL, Bonomo RA, Mathers AJ, van Duin D, Clancy CJ. Infectious Diseases Society of America 2022 Guidance on the Treatment of Extended-Spectrum beta-lactamase Producing Enterobacterales (ESBL-E), Carbapenem-Resistant Enterobacterales (CRE), and Pseudomonas aeruginosa with Difficult-to-Treat Resistance (DTR-P. aeruginosa). Clin Infect Dis. 2022 Aug 25;75(2):187-212. doi: 10.1093/cid/ciac268. PMID 35439291
- [Background] Hu F, Guo Y, Yang Y, Zheng Y, Wu S, Jiang X, Zhu D, Wang F; China Antimicrobial Surveillance Network (CHINET) Study Group. Resistance reported from China antimicrobial surveillance network (CHINET) in 2018. Eur J Clin Microbiol Infect Dis. 2019 Dec;38(12):2275-2281. doi: 10.1007/s10096-019-03673-1. Epub 2019 Sep 2. PMID 31478103
- [Background] Karlowsky JA, Lob SH, Kazmierczak KM, Young K, Motyl MR, Sahm DF. In-vitro activity of imipenem/relebactam and key beta-lactam agents against Gram-negative bacilli isolated from lower respiratory tract infection samples of intensive care unit patients - SMART Surveillance United States 2015-2017. Int J Antimicrob Agents. 2020 Jan;55(1):105841. doi: 10.1016/j.ijantimicag.2019.10.022. Epub 2019 Nov 6. PMID 31704217
- [Background] Rosenthal VD, Bat-Erdene I, Gupta D, Belkebir S, Rajhans P, Zand F, Myatra SN, Afeef M, Tanzi VL, Muralidharan S, Gurskis V, Al-Abdely HM, El-Kholy A, AlKhawaja SAA, Sen S, Mehta Y, Rai V, Hung NV, Sayed AF, Guerrero-Toapanta FM, Elahi N, Morfin-Otero MDR, Somabutr S, De-Carvalho BM, Magdarao MS, Velinova VA, Quesada-Mora AM, Anguseva T, Ikram A, Aguilar-de-Moros D, Duszynska W, Mejia N, Horhat FG, Belskiy V, Mioljevic V, Di-Silvestre G, Furova K, Gamar-Elanbya MO, Gupta U, Abidi K, Raka L, Guo X, Luque-Torres MT, Jayatilleke K, Ben-Jaballah N, Gikas A, Sandoval-Castillo HR, Trotter A, Valderrama-Beltran SL, Leblebicioglu H; International Nosocomial Infection Control Consortium. International Nosocomial Infection Control Consortium (INICC) report, data summary of 45 countries for 2012-2017: Device-associated module. Am J Infect Control. 2020 Apr;48(4):423-432. doi: 10.1016/j.ajic.2019.08.023. Epub 2019 Oct 29. PMID 31676155
- [Background] Sader HS, Streit JM, Carvalhaes CG, Huband MD, Shortridge D, Mendes RE, Castanheira M. Frequency of occurrence and antimicrobial susceptibility of bacteria isolated from respiratory samples of patients hospitalized with pneumonia in Western Europe, Eastern Europe and the USA: results from the SENTRY Antimicrobial Surveillance Program (2016-19). JAC Antimicrob Resist. 2021 Sep 2;3(3):dlab117. doi: 10.1093/jacamr/dlab117. eCollection 2021 Sep. PMID 34671728
- [Background] Hu F, Yuan L, Yang Y, Xu Y, Huang Y, Hu Y, Ai X, Zhuo C, Su D, Shan B, Du Y, Yu Y, Lin J, Sun Z, Chen Z, Xu Y, Zhang X, Wang C, He L, Ni Y, Zhang Y, Lin D, Zhu D, Zhang Y. A multicenter investigation of 2,773 cases of bloodstream infections based on China antimicrobial surveillance network (CHINET). Front Cell Infect Microbiol. 2022 Dec 15;12:1075185. doi: 10.3389/fcimb.2022.1075185. eCollection 2022. PMID 36590586
- [Background] Tabah A, Buetti N, Staiquly Q, Ruckly S, Akova M, Aslan AT, Leone M, Conway Morris A, Bassetti M, Arvaniti K, Lipman J, Ferrer R, Qiu H, Paiva JA, Povoa P, De Bus L, De Waele J, Zand F, Gurjar M, Alsisi A, Abidi K, Bracht H, Hayashi Y, Jeon K, Elhadi M, Barbier F, Timsit JF; EUROBACT-2 Study Group, ESICM, ESCMID ESGCIP and the OUTCOMEREA Network. Epidemiology and outcomes of hospital-acquired bloodstream infections in intensive care unit patients: the EUROBACT-2 international cohort study. Intensive Care Med. 2023 Feb;49(2):178-190. doi: 10.1007/s00134-022-06944-2. Epub 2023 Feb 10. PMID 36764959